CLINICAL TRIAL: NCT03940209
Title: Addressing Basic Needs to Improve Diabetes Outcomes in Medicaid Beneficiaries
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Louisiana Healthcare Connections (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HRPO201811020; 1R01DK115916-01A1 (NIH)
Record Dates: First submitted 2019-05-01; First posted 2019-05-07 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Low Income Population; Diabetes Mellitus, Type 2; Pragmatic clinical trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: In a pragmatic randomized trial, eligible participants who complete a baseline assessment will be randomly assigned to either a basic needs navigation intervention or usual care.
Who Masked: Investigator
Masking Description: Survey administrators also will be blinded to individual participant's study group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Medicaid beneficiaries in this arm will have all the usual resources available to them through their health plan including access to a physician network, case management resources, and other educational and health-focused resources and activities.
- Basic needs navigation (Experimental): Medicaid beneficiaries in this arm will have all the usual resources available to them through their health plan (usual care) as well as a navigator for 6 months to address any unmet basic needs, provide instrumental and emotional social support, and improve self-management capabilities.
  Interventions: Behavioral: Basic needs navigation

INTERVENTIONS:
Behavioral: Basic needs navigation — Navigators will help participants address unmet basic needs for 6 months by telephone. Either party can initiate a call. On every call, navigators will: (1) review unmet needs previously reported (baseline survey for first call) and ask participants to report new needs; (2) jointly prioritize among multiple needs based on severity and resource availability; (3) identify community resources that could help solve the problem; (4) evaluate eligibility for those resources; and (5) prepare participants to interact with service agencies and/or act as an advocate on their behalf. On each subsequent call, navigators will review progress toward resolving those needs, assess emergent needs, and adapt priorities accordingly. Navigators will provide instrumental and emotional social support through regular friendly contact, and will attempt to reduce barriers to needs resolution to improve stability and security for participants longer-term.
  Arms: Basic needs navigation

SUMMARY:
This pragmatic randomized trial will test the effectiveness of a basic needs navigation intervention compared to usual care among 500 adults (ages 18-75) with Medicaid, type 2 diabetes, and 1 or more unmet basic needs. Basic needs includes having such things as adequate food, housing, personal safety, and money for necessities. The primary study hypothesis is that participants who receive navigation to address unmet basic needs will have a greater reduction (M=0.5%) in HbA1c pre-post compared with participants receiving usual care. Consistent with the study's conceptual model, the effects of unmet basic needs on barriers to self-care (e.g., attention, stress, sleep), health behaviors (e.g., glucose monitoring, diet, clinical screenings) and health outcomes (e.g., emergency department utilization, hospitalization, quality of life) will be examined.

DETAILED DESCRIPTION:
Type 2 diabetes affects over 29 million US adults, with a disproportionate burden of disease borne by low-income populations. Effective self-management requires attention, planning, follow-through and consistent performance of multiple health behaviors to prevent negative health outcomes. For low-income individuals, though, health improvement is often superseded by the drive to fulfill basic needs such as food, housing, personal safety, and money for necessities. Having unmet basic needs can overwhelm a person's ability to maintain health behaviors. Prior research has demonstrated that with more unmet basic needs, low-income individuals are less likely to even remember or act on a referral for needed health services. However, when unmet needs are resolved and/or people have a personal navigator to help, the likelihood of acting on a health referral significantly increases. Traditionally, patient navigators help coordinate care, manage disease or promote screening and preventive behaviors. This study will expand the role of navigators to include identifying and resolving unmet basic needs, which is expected to facilitate behavior change and improve health outcomes. This approach will be tested in a pragmatic randomized trial conducted in partnership with Louisiana Healthcare Connections, the largest Medicaid managed care plan in Louisiana. This study will test the effectiveness of a basic needs navigation intervention compared to usual care among 500 adults (ages 18-75) with Medicaid, type 2 diabetes, and 1 or more unmet basic needs. The primary hypothesis is that intervention participants will have a greater reduction (M=0.5%) in HbA1c pre-post compared with usual care participants. Consistent with the study's conceptual model, the effects of unmet basic needs on barriers to self-care (e.g., attention, stress, sleep), health behaviors (e.g., glucose monitoring, diet, clinical screenings) and health outcomes (e.g., emergency department utilization, hospitalization, quality of life) will be examined. Louisiana Healthcare Connections will identify eligible members for study recruitment and provide basic needs navigation for 6 months. The research team will recruit, enroll, randomize, and survey study participants by phone at baseline and 3-, 6- and 12-month follow up. HbA1c data will be obtained from electronic medical records to assess change.

ELIGIBILITY:
Inclusion Criteria:

* Medicaid beneficiary
* Member of Louisiana Healthcare Connections
* Age 18-75 years old
* Diagnosed with type 2 diabetes
* Had a HbA1c test in the 3-4 months prior to baseline assessment

Exclusion Criteria:

* HbA1c <7.0 in the 3-4 months prior to baseline assessment
* Enrolled in case management at Louisiana Healthcare Connections in the 3 months prior to baseline assessment
* Are currently pregnant or have only been diagnosed with gestational diabetes at baseline
* Have cognitive or hearing impairments that significantly impede participation in telephone-based survey and intervention protocols.
* Individuals not living independently (e.g., nursing homes, rehab or correctional facilities)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 12 months
  Glycated haemoglobin (A1c) values will be abstracted from participants' medical record lab reports reflect average plasma glucose concentration over 8-12 weeks

SECONDARY OUTCOMES:
Health-related Quality of Life | 12 months
  Physical and mental summary (subscale) scores from the Short Form-12 item (SF-12) self-report survey instrument will be created following standard scoring guides. Responses are weighted (using regression weights from a general United States population) then summed then standardized to a mean of 50 and standard deviation of 10 (Range 0-100). Higher scores indicate better health status and better health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Investigators may contact study Principal Investigators and complete a data sharing agreement.

REFERENCES:
- [Background] Kreuter MW, McQueen A, Boyum S, Fu Q. Unmet basic needs and health intervention effectiveness in low-income populations. Prev Med. 2016 Oct;91:70-75. doi: 10.1016/j.ypmed.2016.08.006. Epub 2016 Aug 3. PMID 27496395
- [Background] Thompson T, McQueen A, Croston M, Luke A, Caito N, Quinn K, Funaro J, Kreuter MW. Social Needs and Health-Related Outcomes Among Medicaid Beneficiaries. Health Educ Behav. 2019 Jun;46(3):436-444. doi: 10.1177/1090198118822724. Epub 2019 Jan 17. PMID 30654655
- [Background] McQueen A, Roberts C, Garg R, Caburnay C, Fu Q, Gordon J, Bush T, Pokojski R, Thompson T, Kreuter M. Specialized tobacco quitline and basic needs navigation interventions to increase cessation among low income smokers: Study protocol for a randomized controlled trial. Contemp Clin Trials. 2019 May;80:40-47. doi: 10.1016/j.cct.2019.03.009. Epub 2019 Mar 20. PMID 30904596